CLINICAL TRIAL: NCT04815772
Title: Evaluation of Diabetes Mellitus and Smoking on Periodontitis Classifications Using the 1999 and 2018 Periodontal Disease Classifications: a Retrospective Study
Brief Title: Evaluation of the 1999 and 2018 Periodontal Disease Classifications: a Retrospective Study
Status: Completed | Type: Observational
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Ekin Besiroglu, associate professor, Okan University
Other Study IDs: 56665618-204.01.07-22
Record Dates: First submitted 2021-03-19; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus; Smoking; Periodontal Diseases
MeSH Terms: conditions — Diabetes Mellitus; Smoking; Periodontal Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of present study was to evaluate how the 2018 classification reflects the severity, extent and progression of the disease, taking into account the risk factors for periodontal disease, smoking and diabetes, when compared with the 1999 classification.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a complete periodontal chart and full mouth radiographic series at baseline
* Diabetes Mellitus:Patients who consulted by an internist/endocrinologist and underwent HbA1c measurements in the last three months.
* Smoking status:All current smokers who had smoked more than 100 cigarettes in their lifetimes and used cigarettes for more than five years
* Patients meeting the case definition of periodontitis
* Relative radiographic bone loss(in %) was assessed on peri-apical radiograph films

Exclusion Criteria:

* individuals with a systemic disease other than diabetes
* Smokers not reporting the number of cigarette/days or patient(s) with diabetes that do not report Hemoglobin A1c (HbA1c) test results for diabetes.
* individuals who do not suffer from periodontitis
* Patients with inaccessible files because of bad debt, destroyed record, or deceased.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The individuals with periodontitis who participated in the study were evaluated in three categories:
  * individuals who do not smoke and do not have any illnesses
  * non-smoking individuals with diabetes
  * individuals who smoke and have no systemic disease
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
The advantages of including the effect of diabetes and smoking on periodontal disease in the 2018 classification compared to the 1999 classification | The present retrospective study included individuals who were examined and had periodontal measurements made and recorded at the Istanbul Okan University Periodontology Department between 09/01/2018 and 12/01/2019.
  In our study, both classifications reflected the severity of periodontal disease differently. The 2018 classification outperformed the 1999 classification for staging and grading of periodontitis severity and progression. Consideration of the risk factors listed in the 2018 classification has been useful approach for correct diagnosis, evidence-based clinical decisions, prognosis of treatment, and periodontal disease prevention. The 2018 periodontal disease classification is more detailed and comprehensive than the 1999 classification, and this classification is thought to revise the criticisms of the 1999 classification.

CONTACTS AND LOCATIONS:
Overall Officials: ekin Beşiroğlu, 1, Study Director — Okan University
Locations (1):
- İstanbul Okan University, Istanbul, Turkey (Türkiye)